CLINICAL TRIAL: NCT00421772
Title: Prospective Follow-up of a Multicentric Cohort of Children With Prenatal Discovery of Mild Isolated Cerebral Ventriculomegaly. Evaluation at 2 and 5 Years.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Other Study IDs: PHRC-05-03; DGS : 2006/0432; CCPPRB : 2006/08
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2007-01

CONDITIONS: Cerebral Ventriculomegaly
Keywords: cerebral ventriculomegaly; prenatal diagnostic; neuropsychological outcome
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Isolated uni or bilateral mild cerebral ventriculomegaly represents the most frequent "minor" cerebral anomalies discovered by antenatal echography. There are not French data making it possible to specify the incidence and the prevalence of this pathology and international data of the prevalence are very heterogeneous, going, according to the published series, of 1.48 to 22 per 1000 births.

The prognostic of ventriculomegaly remains dubious : the studies have small populations, are for the majority retrospectives with a short and often vague follow-up. The announced rate of after-effects varies between 0 and 48 %.

The objective of this study is to evaluate the neuropsychological development until the 5 years age of the children for whom a prenatally diagnosis of mild isolated ventriculomegaly was carried (absence of another cerebral or extra-cerebral anomaly in imagery and a negative aetiology). This prospective cohort will be compared with children for whom no neurological anomaly was prenatally detected.

The children diagnosed for an mild isolated cerebral ventriculomegaly will be identified by the investigators among medical files of the Centers of Prenatal Diagnosis (CPDPN) of the UH of Angers and the UH of Nantes. The patient inclusion will be done at the 2 years age after parental agreement, with a follow-up at 5 years. The control children will be included under the same conditions after having ensured of the normality of the echographies of 22 and 30 gestational weeks. The follow-up of these 2 cohorts will be based on the 2 years obligatory paediatric examination, and on the network "Naitre ensemble" set up in the Pays de la Loire Loire. In addition to the clinical routine examinations, standardized neuropsychological examinations will be done (Brunet Lezine Revised score at 2 years, NEPSY at 5 years and ASQ at 2 and 5 years).

This study will allow to compare the neuropsychological development at school age of the children diagnosed for a foetal mild, apparently isolated, cerebral ventriculomegaly from children not presenting any foetal anomaly, to evaluate the incidence of the mild isolated ventriculomegaly, to identify the predictive factors of the neuropsychological anomalies in the children diagnosed for ventriculomegaly and to compare (in the children diagnosed for ventriculomegaly), the neuropsychological development at the school age of the children having a ventricular atrium between 10 and 12 mm with those having a ventricular atrium between 12,1 and 15 mm.

This study will allow to define the neuropsychological morbidity of the foetal mild isolated cerebral ventriculomegaly and will allow to define the best clinical and educational follow up of these children and their family.

ELIGIBILITY:
Inclusion criteria : case children

* Written informed consent
* Diagnosis of foetal mild isolated cerebral ventriculomegaly at 32 gestational weeks by the Centers of Prenatal Diagnosis (CPDPN) of the UH of Angers and the UH of Nantes
* Age : 22 to 26 months

Inclusion criteria : control children

* Written informed consent
* Negative diagnostic of foetal cerebral ventriculomegaly at the prenatal echography made at 22 gestational weeks
* Age : 22 to 26 months

Non-inclusion criteria : case children

* Preterm birth (< 37 weeks of gestation)
* APGAR ≤ 3 at 5 minutes after birth
* Serious prenatal pathology with neurologic aspect requing intensive care
* postnatal hydrocephalus
* Diagnostic of a eurological pathology at birth
* Diagnostic d'une pathologie neurologique associée à la naissance

Non-inclusion criteria : control children

* Preterm birth (< 37 weeks of gestation)
* APGAR ≤ 3 at 5 minutes after birth
* Serious prenatal pathology with neurologic aspect requing intensive care
* postnatal hydrocephalus
* Diagnostic of a neurological pathology at birth
* Cerebral or extracerebral anomaly at the prenatal echographies
* Chromosomal anomaly discovered after birth

Ages: 22 Months to 26 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 245
Dates: Start 2007-01; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Claude BOUDERLIQUE, MD, Principal Investigator — UH of Angers
Locations (2):
- France (2):
  - UH of Angers, Angers
  - UH of Nantes, Nantes